CLINICAL TRIAL: NCT01816646
Title: Intravesical Cidofovir Instillation in HSCT Recipients With Hemorrhagic Cystitis: A Single Dose Pharmacokinetic Study
Brief Title: Intravesical Cidofovir for Hemorrhagic Cystitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0903; NCI-2013-02184 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Blood And Marrow Transplantation
Keywords: Blood And Marrow Transplantation; Hemorrhagic Cystitis; Bleeding from bladder; Foley catheter; Probenecid; Cidofovir; Vistide
MeSH Terms: conditions — Cystitis, Hemorrhagic | interventions — Cidofovir; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cidofovir (Experimental): Patients receive a single dose of 2.5 mg/kg of cidofovir administered in 100 ml of normal saline solution through a transurethral catheter inside the bladder. The urinary catheter will be clamped for 2 hours. Probenecid 2 grams by mouth given approximately 3 hours prior to the bladder instillation of cidofovir.
  Interventions: Drug: Cidofovir; Drug: Probenecid

INTERVENTIONS:
Drug: Cidofovir — 2.5 mg/kg of cidofovir administered in 100 ml of normal saline solution through a transurethral catheter inside the bladder. The urinary catheter will be clamped for 2 hours.
  Other Names: Vistide
Drug: Probenecid — 2 grams by mouth given approximately 3 hours prior to the bladder instillation of cidofovir.

SUMMARY:
The goal of this clinical research study is to learn how the drug cidofovir given as 1 dose directly into the bladder is absorbed by the body. Researchers also want to measure the amount of study drug in the body at different time points. The safety and tolerability of this drug will also be studied.

Cidofovir is designed to fight certain viruses by blocking the virus cells from dividing.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, on Day 1, you may receive some fluid for hydration by vein and then cidofovir will be put into your bladder through your foley catheter. The catheter will be clamped shut for 2 hours to keep the drug inside your bladder. After 2 hours, the catheter will be unclamped so that the drug may drain out. If you were receiving bladder irrigation (where the bladder is flushed with water) as therapy for hemorrhagic cystitis, this therapy will be restarted after your dose of cidofovir.

Pharmacokinetic (PK) Testing:

On Day 1, blood (about 2 teaspoons each time) will be drawn for PK testing approximately 1 hour (+/- 15 minutes) before the dose, and then again at 1 hour (+/- 15 minutes), 2 hours (+/- 15 minutes), 4 hours (+/- 1 hour), 14 hours (+/- 1 hour) and 24 hours (+/- 1 hour) after the dose. A PK sample will also be drawn on Day 14 (+- 2 days) after the dose. PK testing measures the amount of study drug in the body at different time points.

Virus Testing:

During this study, urine and blood will be collected and used for research to test for certain viruses, including the type of infection you had when you joined this study.

Before and after the cidofovir dose on Day 1, Day 3 (+/- 1 day), Day 7 (+/- 2 days) and again on Day 14 (+/- 2 days) urine and blood (about 1 teaspoon) will be collected for virus testing.

Length of Study Participation:

Your active study participation will be over after the Day 30 follow-up phone call (below). If you experienced a side effect, the study staff will continue checking your medical records until the side effect becomes stable or gets better.

Follow-Up:

On Day 3 (+/- 1 day):

* You will have a physical exam.
* Your vital signs will be measured, and you will be asked about any symptoms you may be having.
* Urine will be collected for routine tests
* Blood (about 1 teaspoon) will be drawn for routine tests.

On Day 7 (+/- 2 days):

* You will have a physical exam.
* Your vital signs will be measured, and you will be asked about any symptoms you may be having.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Urine will be collected for routine tests.

On Day 14 (+/- 2 days):

* You will be asked about any symptoms you may be having.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Urine will be collected for routine tests.

On Day 30 (+/- 2 days), you will be contacted by phone and asked about any side effects you may be having. This call will take about 10 minutes.

This is an investigational study. Cidofovir given by injection is commercially available and FDA approved to treat CMV in patients with HIV. Its use in this study is investigational.

Up to 6 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Polyoma BK or adenovirus viruria has been established either by positive urine cytology or by PCR for BK virus or by positive urine culture for adenovirus.
2. The patient has either gross hematuria and/or passes blood clots.
3. Signed informed consent form containing all potential serious adverse events related to cidofovir use as given on the package insert.
4. Hospitalized patients with a Foley catheter.
5. Women of childbearing potential (Women who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy) must agree to use 2 acceptable methods of birth control (e. g., barrier method (such and condom or diaphragm) and another form, such as an intrauterine device (IUD) or hormonal birth control, during the study period and for a period of 2 months afterward. Males must also agree to use an acceptable method of birth control (barrier method) during the study period and for 2 months afterward.

Exclusion Criteria:

1. Serum creatinine >2 mg/dl and/or calculated creatinine clearance < 50 ml/min using the Cockcroft-Gault Creatinine Clearance formula (CrCl). CrCl = {(140-Age) x Weight (kgs) x 0.85 (if female)}/ {72x Serum Creatinine (mg/dl)}
2. Urine protein > 100 mg/dl (equivalent to > 2+ proteinuria)
3. Age less than 18 years.
4. Prior therapy with formalin or carboprost 1 mg/dL administered intravesically.
5. Hypersensitivity to cidofovir, probenecid or sulfa-containing medications
6. Patients who have received prior cidofovir therapy within 2 weeks
7. Prior enrollment in the study
8. Women who are pregnant or breast-feeding
9. Evidence of end-organ adenoviral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Systemic Absorption of Cidofovir | 7 days
  Systemic absorption of drug evaluated during and after intravesical administration. Blood collected for each sample in the following schedule:
  1. T0 (pre-instillation)
  2. 1 hour (after instillation)
  3. 2 hours (after instillation-at the time of de-clamping)
  4. 4 hours +/- 1 hour (after instillation)
  5. 14 hours +/- 1 hour (14 hours after instillation or 12 hours from de-clamping).
  6. 24 hours +/- 1 hour after instillation to ensure complete characterization of cidofovir elimination.

CONTACTS AND LOCATIONS:
Overall Officials: Roy F. Chemaly, MD, MPH, MBA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Aitken SL, Zhou J, Ghantoji SS, Kontoyiannis DP, Jones RB, Tam VH, Chemaly RF. Pharmacokinetics and safety of intravesicular cidofovir in allogeneic HSCT recipients. J Antimicrob Chemother. 2016 Mar;71(3):727-30. doi: 10.1093/jac/dkv393. Epub 2015 Nov 26. PMID 26612873
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org